CLINICAL TRIAL: NCT00179803
Title: Phase II Prospective Study of Sequential Myeloablative Chemotherapy With Stem Cell Rescue for the Treatment of Selected High Risk CNS Tumors and Recurrent CNS Tumors
Brief Title: Stem Cell Transplant for High Risk Central Nervous System (CNS) Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stewart Goldman, Attending Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 0398
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Glioblastoma; Astrocytoma; Pineoblastoma; Rhabdoid Tumor; Supratentorial Neoplasms
Keywords: brain tumor; medulloblastoma; germ cell tumor; CNS tumor; glioblastoma; astrocytoma; pineoblastoma; rhabdoid tumor; supratentorial PNET; high grade astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Pinealoma; Rhabdoid Tumor; Supratentorial Neoplasms; Brain Neoplasms; Medulloblastoma; Neoplasms, Germ Cell and Embryonal; Central Nervous System Neoplasms | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: high dose chemotherapy with stem cell rescue thiotepa, carboplatin & etoposide
Oversight: Data Monitoring Committee: No

ARMS (1):
- high dose chemotherapy (Experimental)
  Interventions: Procedure: Stem Cell Transplant

INTERVENTIONS:
Procedure: Stem Cell Transplant — Group A: recurrent medulloblastoma, recurrent germ cell tumor
  * Cytoxan treatment
  * Stem cell autologous harvest
  Group B: GBM, high grade astrocytoma, rhabdoid tumors, pineoblastoma, or supratentorial PNET
  * Carboplatin and Etoposide treatment
  * Autologous stem cell harvest
  The preparatory regimen used for Stem Cell Rescue #1 will be Carboplatinum, VP-16 and Thiotepa. If the patient has recuperated his ANC to >1,000 within 50 days after Stem Cell Rescue #1, (sustained without G-CSF support) a neuroradiographic evaluation will be performed. If there is lack of progression, the patient will then proceed to Stem Cell Rescue # 2 with Cyclophosphamide and Melphalan, followed by stem cell rescue.

SUMMARY:
The primary goal of this study is to determine if a stem cell transplant in patients with newly diagnosed high risk CNS tumors (glioblastoma multiforme [GBM], high grade astrocytoma, pineoblastoma, rhabdoid tumor, supratentorial primitive neuroectodermal tumor [PNET]) increases overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age must be greater than (>) 18 months and less than or equal to (≤) 25 years at the time of diagnosis or recurrence.
* Neuroradiographic evidence of a recurrent posterior fossa medulloblastoma or recurrent CNS germ cell tumor.
* The presence of a histologically confirmed high grade astrocytoma, GBM, rhabdoid tumor, supratentorial PNET, or pineoblastoma either at the time of diagnosis or recurrence.
* Patients must be brought to state of minimum residual disease by surgical reduction and/or chemotherapy and/or radiation therapy or a combination of above prior to myeloablative chemotherapy and tandem stem cell rescue.
* Documentation of chemotherapy sensitivity is required for enrollment. Chemotherapy-sensitive tumors are defined as those tumors which have had a reduction of 50% after 2-4 cycles of chemotherapy (CTX or platinum). For patients with no evidence of disease post resection, continued complete remission after 2-4 cycles of chemotherapy defines chemosensitivity.
* Adequate physiologic function, defined as follows:

  * creatinine clearance > 70 ml/minutes/1.73 m2.
  * SGPT < 10 x normal and bilirubin < 10 mg/dl.
* Adequate complete blood count (CBC): hemoglobin > 10 gm/dl, absolute neutrophil count (ANC) > 1500/ul, and platelets > 100,000/ul.
* Informed consent. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained, in accordance with institutional policies provided by the United States (U.S.) Department of Health and Human Services.
* Protocol approval. Approval for the use of this institution's Human Rights Committee must be obtained in accordance with the institutional assurance policies of the U. S. Department of Health and Human Services.
* Patients with high-risk medulloblastoma after initial surgery.
* To allow non-English speaking patients to participate in this study, bilingual health care services will be provided in the appropriate language.

Exclusion Criteria:

* Patients with brain stem glioma are ineligible.

Ages: 18 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 1998-03; Primary Completion 2008-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine if the use of sequential myeloablative chemotherapy with peripheral blood stem cell rescue will increase the overall survival rate in patients with newly diagnosed high risk CNS tumors | To end of study

SECONDARY OUTCOMES:
The overall survival and progression free survival in children with recurrent CNS malignancies after obtaining a state of minimum residual disease with submyeloablative chemotherapy, surgery, and/or radiation. | To end of study
To determine the progression free survival and overall survival using sequential myeloablative chemotherapy as compared to historical controls with single autologous stem cell rescue following myeloablative chemotherapy. | To end of study
Determine the long term neurocognitive, endocrinologic, cardiopulmonary, and hematologic sequelae of sequential myeloablative chemotherapy and stem cell rescues in patients treated for high risk CNS and recurrent CNS tumors. | To end of study
Determine the feasibility and utility of the myeloablative preparatory regimen of Carboplatinum, VP-16 and Thiotepa administered in an outpatient setting, and to determine the cost savings obtained via this strategy. | To end of study

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States